CLINICAL TRIAL: NCT04492553
Title: Gonadal Dysfunction in Male Long-term Survivors of Malignant Lymphoma; A Prospective Non Randomised Open Label Multicenter Phase Two Study in Male Longterm Survivors of Malignant Lymphoma (Vitality)
Brief Title: Gonadal Dysfunction in Male Long-term Survivors of Malignant Lymphoma; Vitality
Acronym: Vitality
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lars Møller Pedersen (Other)
Collaborators: Besins Healthcare (Industry); Copenhagen University Hospital at Herlev (Other); Zealand University Hospital (Other)
Responsible Party: Sponsor-Investigator, Lars Møller Pedersen, Senior consultant, Herlev Hospital
Organization: Herlev Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Vitality
Record Dates: First submitted 2020-07-27; First posted 2020-07-30 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Hypogonadism
Keywords: quality of life; sexuality; sexual health; EORTC; QLQ-C30; SHQ-22; IIEF-5; hypogonadism; testosterone; cancer; lymphoma; diffuse large b-cell lymphoma; hodgkin
MeSH Terms: conditions — Hypogonadism; Sexuality; Neoplasms; Lymphoma; Lymphoma, Large B-Cell, Diffuse | interventions — Testosterone

STUDY DESIGN:
Intervention Model Description: Cured lymphoma patients who suffer from hypogonadism identified in a previous study, Vitality-Obs, will be treated with testosterone replacement therapy for the duration of one year. Patients are treated after standard indication and in standard doses. All will receive the same treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Testogel (Experimental): All patients will be treated with Testogel. Starting dose is 1 sachet of gel daily applied to the skin of arms, thighs or abdomen. Dose adjustments are made after serum-levels of testosterone. All patients will be treated for a total of 52 weeks, unless they exit the study early because of side-effects or other reasons.
  Interventions: Drug: AndroGel

INTERVENTIONS:
Drug: AndroGel — Treatment indication: hypogonadism after cancer treatment. Dosage: 1-2 sachets a day. Follows standard treatment.
  Other Names: Testogel

SUMMARY:
This study is a prospective non-randomised open label multicenter phase two study in male long-term survivors of malignant lymphoma including Hodgkin Lymphoma (HL) and Diffuse Large B-Cell Lymphoma (DLBCL). The study aims to assess whether low levels of testosterone in the blood of patients cured for aggressive lymphoma, can be effectively treated with Testosterone gel, and if treatment with testosterone can improve their general quality of life. The investigators hypothesize that patients will develop sexual dysfunction and poor quality of life when suffering from untreated reduced level of testosterone.

Cancer treatment is increasingly effective and the overall survival higher, which makes issues like sexuality and long-term quality of life more and more important to address in cured cancer patients. Patient sexuality and quality of life is measured by three questionnaires, and serum testosterone level, during one year of treatment with Testogel. The intention is to show that future follow-up visits should include focus on sexuality and serum testosterone, so relevant patients can be identified and treated for their hormonedeficiency without delay. The expected follow-up program include questionnaires and blood samples, which are easily implemented and without great cost.

DETAILED DESCRIPTION:
Diffuse large B-cell lymphoma and Hodgkin Lymphoma are two aggressive lymphomas often treated with doxorubicin containing chemotherapy. Doxorubicin is an anthracycline and is known to be toxic to both Leydig Cells of the testes and hormone-producing cells of the hypothalamus. Therefore, patients treated with this drug are at risk of developing hypogonadism. Standard follow-up programs do not include analysis of hormone levels or treatment of hypogonadism. With this study the aim is to investigate the effect and toxicity of treatment with exogenous testosterone in male long-term survivors of malignant lymphoma, to clarify whether it is relevant to include serum testosterone and potentially testosterone replacement therapy in standard follow-up programs.

Our Hypothesis:

Hypothesis 1: A significant proportion of long-term male survivors of HL and DLBCL have impaired quality of life (QoL) due to sexual dysfunction.

Hypothesis 2: A significant proportion of long-term male survivors of HL and DLBCL have reduced levels of testosterone.

Hypothesis 3: A significant relationship between QoL, sexual dysfunction and testosterone levels exists.

Hypothesis 4: Substitution with testosterone in carefully selected subgroups will improve sexual function and QoL.

Hypothesis 5: Treatment with testosterone in this setting is safe with acceptable toxicity.

To assess efficacy and safety of treatment with testosterone replacement therapy on hypogonadism in lymphoma patients, blood tests and questionnaires are completed throughout one year of treatment. To assess patient sexuality and quality of life, 3 questionnaires are included; the European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire Core 30 (QLQ C30) for general quality of life, EORTC Sexual Health Questionnaire 22 (SHQ-22) for sexual health and International index of erectile function with 5 questions (IIEF-5) for sexual function.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years at inclusion
2. Male
3. Verified diagnosis of de novo DLBCL or classical HL diagnosed between April 2008 and April 2018 according to World Health Organization (WHO) classification.
4. Completed curative intent first line treatment with anthracycline-containing chemotherapy with or without consolidating radiotherapy, with disease in complete remission at End of Treatment (EOT) Positron Emissions Tomography / Computerized Tomography (PET/CT) at least one year prior to inclusion.
5. Literate in Danish
6. Serum testosterone level below threshold for age adjusted reference level used in the local laboratory at the time of inclusion.

Exclusion Criteria:

1. Concurrent low-grade lymphoma
2. Current or prior lymphoproliferative disease of the central nervous system (CNS)
3. Current or prior lymphoproliferative disease of the testes
4. Contraindications for the treatment with testosterone: Verified prostate cancer / Prostate Specific Antigen (PSA) > 3 ng/ml, cancer of the mammae, primary liver cancer or polycythaemia vera / Hct > 0,49.
5. Mental or physical conditions that are expected to prevent the necessary "compliance" and/or "adherence" in relation to the study procedures
6. Current or prior anabolic steroid drug abuse
7. Treatment with second line chemotherapy or high dose therapy.
8. Known allergies to additives in Testogel.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Gender is based on social security number
Enrollment: 7 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-11-10 (Actual); Study Completion 2022-11-10 (Actual)

PRIMARY OUTCOMES:
Effect of testosterone on QLQ C-30 score | 1 year
  Effect of treatment with testosterone on QLQ C30 score from baseline to end of study (12 months after inclusion). Scores a measured from 3 scales; function, symptoms and global health. Highest score is 100. Scoring after an algorithm.

SECONDARY OUTCOMES:
Effect of testosterone on QLQ SHQ-22 score | 1 year
  Effect of treatment with testosterone on QLQ SHQ-22 score from baseline to end of study (12 months after inclusion). Scores a measured from 2 scales; function and symptoms. Highest score is 100. Scoring after an algorithm.
Effect of testosterone on IIEF-5 score | 1 year
  Effect of treatment with testosterone on symptoms of hypogonadism (IIEF-5 score) from baseline to end of study (12 months after inclusion). IIEF-5 is based on 5 questions. Scores range from 5 to 25, Lower scores mean higher degree of erectile dysfunction.
Time from baseline until significant change in questionnaire scores are seen | 1 year
  Time from baseline to a significant decrease in QLQ C30, QLQ SHQ-22 (a little change 5-10 points difference, moderate change 10-20, very much change above 20) and IIEF-5 (changing from at least one category to the next) score is seen.
S-testosteron change | 1 year
  S-testosterone from baseline to end of study (12 months after inclusion).
Testosterone dose needed for significant change in scores | 1 year
  Testosterone dose needed before significant decrease in QLQ C30, QLQ SHQ-22 and IIEF-5 score. Dosing range from 1 to 2 sachets of Testogel per day.

CONTACTS AND LOCATIONS:
Overall Officials: Lars Møller Pedersen, MD, Principal Investigator — Zealand University Hospital
Locations (3):
- Denmark (3):
  - Copenhagen University Hospital, Copenhagen
  - Herlev University Hospital, Herlev
  - Zealand University Hospital, Roskilde